CLINICAL TRIAL: NCT02182674
Title: A Randomized, Double Blind, Crossover, Placebo- and Active Controlled Dose Confirmation Study of Combivent HFA Inhalation Aerosol in Patients With COPD
Brief Title: A Confirmation Study of Combivent HFA Inhalation Aerosol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.25
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol, Ipratropium Drug Combination

ARMS (2):
- Combivent HFA (Experimental)
  Interventions: Drug: Placebo Combivent HFA; Drug: Combivent HFA
- Combivent (CFC) (Active Comparator)
  Interventions: Drug: Combivent (CFC); Drug: Placebo Combivent (CFC)

INTERVENTIONS:
Drug: Placebo Combivent HFA
  Arms: Combivent HFA
Drug: Combivent HFA
  Arms: Combivent HFA
Drug: Combivent (CFC)
  Arms: Combivent (CFC)
Drug: Placebo Combivent (CFC)
  Arms: Combivent (CFC)

SUMMARY:
Study to demonstrate the comparability of two puffs of Combivent hydrofluoroalkane (HFA) inhalation aerosol (18 mcg ipratropium bromide/100 mcg albuterol sulfate / per puff) to two puffs of the marketed chlorofluorocarbon (CFC) containing product, Combivent (CFC) inhalation aerosol (18 mcg ipratropium bromide/103 mcg albuterol sulfate / per puff). The dose response profile, safety and pharmacokinetics of Combivent HFA formulation are to be characterized.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were to have a diagnosis of COPD and must have met the following criteria at visit 1: Patients were to have relatively stable, moderate to severe airway obstruction with a baseline forced expiratory volume in one second (FEV1) <=65 % of predicted normal and FEV1 / forced vital capacity (FVC) <=70 %.
2. Patients must have demonstrated a >= 015 % improvement in baseline FEV1 within one hour after the inhalation of two puffs of Combivent (CFC) inhalation aerosol (18 mcg ipratropium bromide/103 mcg albuterol sulfate per actuation; ex-mouthpiece dose)
3. Male or female patients 40 years of age or older.
4. Patients must have had a smoking history of more than ten pack-year. A pack-year is defined as the equivalent of smoking on pack of 20 cigarettes per day for a year.
5. Patients must have been able to perform technical satisfactory pulmonary function test.
6. Patients must have been able to be trained in the proper use of a metered dose inhalator (MDI)
7. All patients must have signed an informed consent form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications.

Exclusion Criteria:

1. Patients with significant disease other than COPD were to be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinical relevant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defined a disease listed as an exclusion criterion, the patient was to be excluded.
3. All patients with a serum glutamic-oxaloacetic transaminase (SGOT) > 80 IU/L, serum glutamic pyruvic transaminase (SGPT) > 80 IU/L, bilirubin > 2.0 mg/dL or creatinine > 2.0 mg/dL were to be excluded regardless of the clinical condition. Repeat laboratory evaluation was not to be conducted in these patients.
4. Patients who had total blood eosinophil count >= 600/mm³. A repeat eosinophil count was not to be conducted in these patients.
5. Patients with a recent history (i.e., one year or less) of myocardial infarction.
6. Patients with a recent history (i.e., three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
7. Patients with a history of cancer, other than treated basal cell carcinoma, within the last five years.
8. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
9. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history or a thoracotomy for other reasons were to be evaluated as per exclusion criteria no. 1.
10. Patients with a history of asthma, allergic rhinitis or atopy.
11. Patients with a history of or active alcohol or drug abuse.
12. Patients with known active tuberculosis.
13. Patients with an upper respiratory tract infection or COPD exacerbation in the six weeks prior to screening visit (Visit 1) or between the screening visit and visit 2.
14. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
15. Patients with known narrow-angle glaucoma.
16. Patients with current significant psychiatric disorder.
17. Patients with regular use of daytime oxygen therapy.
18. Patients who were being treated with beta blocker medication, mono amine oxidase (MAO) inhibitors or tricyclic antidepressants.
19. Patients who were being treated with cromolyn sodium or nedocromil sodium.
20. Patients who were being treated with antihistamines.
21. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose before screening visit or a change between the screening visit and visit 2) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
22. Patients who had been treated with oral beta adrenergics or long-acting beta-adrenergics such as salmeterol (Serevent) and formoterol in the two weeks prior to the screening visit or between the screening visit and visit 2.
23. Patients who have had changes in their therapeutic plan within the last six weeks prior to the screening visit or between the screening visit and visit 2, excluding changes from long acting or oral beta-adrenergics to short acting inhaled beta-adrenergics for purposes of this trial.
24. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception.
25. Patients with known hypersensitivity to anticholinergic or beta-agonist drugs or any other component of either Combivent formulation.
26. Patients who had taken an investigational drug within one month or six half lives (whichever is greater) prior to the screening visit.
27. Previous participation in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2000-10; Primary Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Average forced expiratory volume in the first second (FEV1) response calculated as area under the curve above test-day baseline from time 0 to 6 hours divided by six (AUC0-6h) | 0, 1, 2, 3, 4, 5 and 6 hours post drug administration

SECONDARY OUTCOMES:
onset of therapeutic FEV1 response | up to 8 hours post drug administration
peak FEV1 | up to 8 hours post drug administration
time to peak FEV1 | up to 8 hours post drug administration
average of FEV1, pictured as area under the curve (AUC0-8h) | 0, 1, 2, 3, 4, 5, 6 and 8 hours post drug administration
individual FEV1 | 0, 1, 2, 3, 4, 5, 6 and 8 hours post drug administration
individual forced vital capacity (FVC) | 0, 1, 2, 3, 4, 5, 6 and 8 hours post drug administration
average of FVC, pictured as area under the curve (AUC0-8h) | 0, 1, 2, 3, 4, 5, 6 and 8 hours post drug administration
peak FVC | up to 8 hours post drug administration
ipratropium plasma concentration | pre-treatment; 5, 15, 30 minutes and 1, 2, 4 and 8 hours post drug administration
albuterol plasma concentration | pre-treatment; 5, 15, 30 minutes and 1, 2, 4 and 8 hours post drug administration
ipratropium amount from renal excretion (Ae0-2, Ae0-8) | pre-treatment, 0 to 2 hours and 2 to 8 hours post drug administration
albuterol amount from renal excretion (Ae0-2, Ae0-8) | pre-treatment, 0 to 2 hours and 2 to 8 hours post drug administration
ipratropium plasma concentration (AUC0-8h) | 5, 15, 30 minutes and 1, 2, 4 and 8 hours post drug administration
albuterol plasma concentration (AUC0-8h) | 5, 15, 30 minutes and 1, 2, 4 and 8 hours post drug administration
number of patients with Adverse Events | up to day 49 after first drug administartion
change from baseline in pulse rate and blood pressure | up to day 49 after first drug administartion
change from baseline in physical examination, laboratory test and 12-lead ECG | up to day 49 after first drug administartion